CLINICAL TRIAL: NCT04959994
Title: Small Bowel Evaluation Using Novel Motorized Spiral Enteroscopy - Prospective Non-controlled Clinical Study From a Single Tertiary Care Centre.
Brief Title: Small Bowel Evaluation Using Novel Motorized Spiral Enteroscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Other Study IDs: AIG/IEC-BH&R 15/06.2021-01
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Small Bowel Disease
Keywords: Small bowel disease; Deep enteroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Novel Motorized Spiral Enteroscopy — All the patients with suspected small bowel disease and an indication to undergo total enteroscopy and satisfying inclusion criteria will undergo novel motorized spiral enteroscopy

SUMMARY:
Small bowel evaluation using Novel Motorized Spiral Enteroscopy - Prospective non-controlled clinical study from a single tertiary care centre.

Data regarding the safety and efficacy of Novel Motorized Spiral Enteroscopy in the evaluation of the small bowel, most of them are retrospective. This study is being planned to collect the data prospectively for all the patients undergoing this procedure at our center including the follow up at 1 month for any adverse events.This will enlighten us in understanding the role of Novel Motorized Spiral in the evaluation of the small bowel Enteroscopy in the small bowel evaluation.

DETAILED DESCRIPTION:
1. Introduction Few studies have been published till now regarding the safety and efficacy of Novel Motorized Spiral Enteroscopy in the evaluation of the small bowel, most of them are retrospective. This study is being planned to collect the data prospectively for all the patients undergoing this procedure at our centre including the follow up at 1 month for any adverse events. This will help us to develop our understanding the role of Novel Motorized Spiral Enteroscopy in the small bowel evaluation.
2. Rationale Prospective study evaluating the efficacy of the Novel Motorized Spiral Enteroscopy is lacking. This study will help in understanding the efficacy and safety of the procedure in the evaluation of the small bowel diseases.
3. Study Population All the patients who will undergo small bowel evaluation using Novel Motorized Spiral Enteroscopy at AIG Hospitals, Gachibowli, Hyderabad, Telangana, India
4. Methodology Patients with suspected small bowel disease with an indication for total enteroscopy will undergo Novel Motorized Spiral Enteroscopy at AIG hospitals. Patient record including the Demographic details, Indications, Pre-Anaesthesia evaluation, History of any previous surgery or prior enteroscopy. Procedure technical success, Total enteroscopic small bowel evaluation rate or extent of examination. Therapeutic procedure underwent, Total Procedure time, Diagnosis, Recovery from anaesthesia time record will be maintained. All the patients will be followed up telephonically for any possible adverse event upto 30 days.

Patient details will be recorded in a proforma after taking proper informed consent.

4a. Inclusion Criteria

1. Patients with small bowel disease with an indication for Motorized spiral enteroscopy
2. Overt or obscure Gastrointestinal bleeding
3. Iron deficiency anaemia
4. Chronic diarrhoea
5. Abdominal pain for evaluation with suspected small bowel involvement.
6. IBD requiring small bowel evaluation
7. Polyposis syndrome requiring small bowel evaluation
8. Small bowel subacute obstruction
9. Refractory celiac disease

4b. Exclusion criteria

1. Weight less than 30 kg
2. Large gastric or oesophageal varices
3. Any medical contraindication to standard enteroscopy
4. Any prior history of gastric , small bowel , large bowel surgery
5. Acute obstruction of small bowel
6. Suspected GI perforation
7. Any contraindication for general anaesthesia
8. Lack of informed consent.

4c. Subject recruitment All the patients who will undergo the procedure according to the inclusion and exclusion criteria will be taken. Prospectively their records will be maintained by proforma at AIG hospitals, Gachibowli.

4d. Randomization and blinding - NIL Single group assignment with no randomization

4e. Method of assessment This will be a non- controlled single group assignment study,All antegrade power spiral enteroscopy procedures will be performed under elective general anesthesia with nasotracheal intubation.Retrograde power spiral enteroscopy procedures will be performed under deep sedation using propofol.A prophylactic wire guided dilatation using Savary - Gilliard dilator up to 20 mm will be done in all the patients. After the maximal depth of insertion via the antegrade route hemoclip or Indiaink will be applied to mark the maximal depth of insertion and retrograde enteroscopy will be done to try to trace the hemoclip on the same or the next day to obtain total enteroscopy.

4f. Stopping or discontinuation criteria- None

5. Sample size calculation All the patients who will undergo Novel Motorized Spiral Enteroscopy will be recorded in a proforma and their follow up at 30 days will be assessed telephonically for a duration of 1 year

6. Statistical analysis The database will be created with Microsoft Excel (Microsoft, Seattle, Wash, USA). Data entry will be done by primary investigator using google forms and it will be stored with the primary investigator. Statistical analyses will be done using SPSS version 25 (IBM Corp., Armonk, NY, USA). Continuous measures will be expressed with sample size, mean (standard deviation), median (range), as and when required. Categorical measures will be presented as number of patients and percentage. The 95% confidence interval will be calculated using exact Clopper-Pearson for diagnostic yield and TER.

7. Ethical justification of the study This is a prospective nonrandomized non-controlled trial with patients not assigned to any specific intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with small bowel disease with an indication for Motorized spiral enteroscopy and age more than 10 years
2. Overt or obscure Gastrointestinal bleeding
3. Iron deficiency anaemia
4. Chronic diarrhoea
5. Abdominal pain for evaluation with suspected small bowel involvement.
6. IBD requiring small bowel evaluation
7. Polyposis syndrome requiring small bowel evaluation
8. Small bowel subacute obstruction
9. Refractory celiac disease

Exclusion Criteria:

1. Weight less than 30 kg
2. Large gastric or oesophageal varices
3. Any medical contraindication to standard enteroscopy
4. Any prior history of gastric , small bowel , large bowel surgery
5. Acute obstruction of small bowel
6. Suspected GI perforation
7. Any contraindication for general anaesthesia
8. Lack of informed consent.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients with suspected small bowel disease satisfying the inclusion criteria and have indications for total enteroscopy will undergo small bowel evaluation using Novel Motorized Spiral Enteroscopy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-06-16 (Estimated); Study Completion 2022-06-16 (Estimated)

PRIMARY OUTCOMES:
Total enteroscopy rate with motorized spiral enteroscopy both via antegrade and the retrograde route. | 2 days
  Rate of examining the total small bowel evaluation using novel motorized spiral enteroscopy

SECONDARY OUTCOMES:
Technical success of antegrade and the retrograde approach | 2 days
  Passage of the scope at least till the duodenojejunal flexure
Total procedural time | 2 days
  Total procedural time beginning from the ligament of trietz to the maximal depth of the insertion via antegrade route and passage of the scope from the ileocecal valve to the maximal depth of the insertion via the retrograde route
Depth of the maximal insertion | 2 days
  Maximal depth of the insertion beyond the ligament of Trietz via the antegrade route and beyond the Ileocecal valve via the retrograde route.
Diagnostic yield | 2 days
  Diagnostic yield, defined as the percentage of procedures with a definitive endoscopic diagnosis (either confirmed a diagnosis from previous imaging or new diagnosis at the anatomic location identified in previous imaging studies).
Therapeutic yield | 2 days
  Therapeutic yield, defined as the percentage of any therapeutic procedures done excluding biopsy and hemoclip application to mark the maximal depth of insertion.
Adverse events | 30 days
  Any adverse events including minor or major which may require surgical intervention or ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Aniruddha P Singh, MBBS,MD,DM, Principal Investigator — AIG hospitals,India; Mohan Ramchandani, MBBS,MD,DM, Study Director — AIG Hospitals,India; Duvur Nageshwar Reddy, Study Chair — AIG Hospitals,India
Locations (1):
- Aniruddha Pratap Singh, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Beyna T, Arvanitakis M, Schneider M, Gerges C, Hoellerich J, Deviere J, Neuhaus H. Total motorized spiral enteroscopy: first prospective clinical feasibility trial. Gastrointest Endosc. 2021 Jun;93(6):1362-1370. doi: 10.1016/j.gie.2020.10.028. Epub 2020 Nov 2. PMID 33144239
- [Result] Beyna T, Arvanitakis M, Schneider M, Gerges C, Boing D, Deviere J, Neuhaus H. Motorised spiral enteroscopy: first prospective clinical feasibility study. Gut. 2021 Feb;70(2):261-267. doi: 10.1136/gutjnl-2019-319908. Epub 2020 Apr 24. PMID 32332141
- [Result] Ramchandani M, Rughwani H, Inavolu P, Singh AP, Tevethia HV, Jagtap N, Sekaran A, Kanakagiri H, Darishetty S, Reddy DN. Diagnostic yield and therapeutic impact of novel motorized spiral enteroscopy in small-bowel disorders: a single-center, real-world experience from a tertiary care hospital (with video). Gastrointest Endosc. 2021 Mar;93(3):616-626. doi: 10.1016/j.gie.2020.07.001. Epub 2020 Jul 12. PMID 32663489